CLINICAL TRIAL: NCT03692780
Title: A Phase I Dose-Finding Followed by Phase IIa Randomized, Double-Blind, Placebo-Controlled, Parallel, Add-on to Cisplatin Plus Docetaxel Study to Evaluate the Safety, Tolerability and Efficacy Profiles of Careseng 1370 to Treat Chemotherapy-Induced Myelosuppression in Advanced Non-Small Cell Lung Cancer (NSCLC) Subjects
Brief Title: Careseng 1370 for Chemotherapy-Induced Myelosuppression
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: At sponsor's discretion
Sponsor: Careseng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Careseng 1370-02
Record Dates: First submitted 2018-09-25; First posted 2018-10-02 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Chemotherapy-Induced Myelosuppression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Careseng 1370 (Experimental)
  Interventions: Drug: Careseng 1370
- Matched Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Careseng 1370 — 4,000mg granules in sachet
  Arms: Careseng 1370
Drug: Placebo — 4,000mg granules in sachet
  Arms: Matched Placebo

SUMMARY:
This is a Phase I/IIa dose-finding (Phase I) followed by randomized, double-blind, placebo-controlled, parallel, add-on to cisplatin + docetaxel (Phase IIa) study to evaluate the safety, tolerability, and efficacy profiles of Careseng 1370 in subjects with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Of either gender aged at least 20 years old
2. Histologically or cytologically confirmed unresectable, locally advanced, metastatic untreated NSCLC and can be accurately assessed by computed tomography/magnetic resonance imaging (CT/MRI) scan (RECIST v1.1) for which regimen of cisplatin + docetaxel is arranged by the investigator; no prior chemotherapy treatment for this disease will be allowed.
3. ECOG performance status score ≤2 and life expectancy ≥12 months
4. Dated and signed informed consent

Exclusion Criteria:

1. Had chemotherapy, therapeutic radiotherapy, or other therapy for NSCLC within 6 weeks before Screening visit
2. Has undergone major surgery within 4 weeks before Screening visit
3. With contraindications to MRI
4. Has elective or planned surgery to be conducted during the trial
5. Has documented brain or leptomeningeal metastases or any cancer other than NSCLC
6. Inadequate hematologic function, as defined by: absolute neutrophil count (ANC) ≤ 1,500/µL; hemoglobin concentration < 10.0 g/dL; and platelet count ≤ 100,000/µL
7. Inadequate hepatic function, as defined by: total bilirubin level > ULN; AST or ALT > 1.5 x ULN; gamma-GT > 2.5 x ULN; ALP > 2.5 x ULN.
8. Inadequate renal function, as defined by: serum creatinine level > 1.5 x ULN; or calculated serum creatinine clearance (Cockcroft-Gault) < 50 mL/min
9. Urinary protein >1+ on dipstick, edema or serum albumin < lower level of normal
10. Any other ≥ grade 3 laboratory abnormality at baseline
11. Inadequate coagulation function, as defined by: INR > 1.5 x ULN or aPTT > 1.5 x ULN
12. Male subject with female spouse/partners who are of childbearing potential refuses to adopt highly effective contraceptives from Screening visit until 7 days after end of study treatment
13. Female subjects with childbearing potential who is pregnant (confirmed by urine or serum pregnancy test) or lactating, refuses to adopt highly effective contraceptives, if heterosexually active, from Screening visit until 7 days after end of study treatment
14. Requirement of anticoagulants, antiplatelet treatments (e.g., warfarin, heparins) from Screening visit until Final visit
15. History of human immunodeficiency virus (HIV) infection
16. Has experienced any grade 3 or 4 gastrointestinal bleeding within 12 weeks before Screening visit
17. Has a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess <6 months before Screening visit, or the subject has a history of poorly controlled or recurrent inflammatory bowel disease (including Crohn's disease or ulcerative colitis)
18. Has participated in a clinical study within 4 weeks prior to Screening visit
19. Has a known allergy to investigational product Careseng 1370, matched placebo, cisplatin, docetaxel or their excipients. If there is suspicion that the subject may have an allergy, the subject should be excluded.
20. Has known alcohol or drug dependency
21. Requirement for ongoing immunosuppressive agents (including azathioprine, mycophenolate, cyclophosphamide, chlorambucil, methotrexate, cyclosporine) or systemic steroid with equivalent dosage higher than prednisolone 30 mg/day for more than 14 days
22. Significant cardiovascular disease, including:

    1. History of New York Heart Association (NYHA) class III or IV congestive heart failure
    2. Ongoing uncontrolled hypertension
    3. History of congenital long QT syndrome
    4. Ongoing prolonged corrected QT (QTc) interval defined as at least 450 msec
    5. History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation)
23. Uncontrolled psychiatric disorder or altered mental status precluding informed consent or necessary testing per investigator's discretion
24. Consumption of herbal preparations/supplements (except for a daily multivitamin/mineral supplement not containing herbal components) within 2 weeks prior to the start of cisplatin + docetaxel or Careseng 1370/matched placebo administration
25. Is not considered to be suitable for this study, in the opinion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Maximum change of absolute neutrophil count (ANC) up to End of Treatment visit | Day 1, 8, 15 22, 29, 36, 43, 50, 57, 64, 71, 78, 85
  End of Treatment will be Day 85

SECONDARY OUTCOMES:
Proportion of subjects with anemia, neutropenia, or thrombocytopenia of all grades at post-treatment visits | Day 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85
Maximum change and by visit change in white blood cell (WBC) count from baseline to post-treatment visits | Day 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85
Maximum change and by visit change in platelet count from baseline to post-treatment visits | Day 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85
Maximum change and by visit change in red blood cell (RBC) count from baseline to post-treatment visits | Day 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85
Maximum change and by visit change in serum C-reactive protein (CRP) level from baseline to post-treatment visits | Day 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85
Maximum change and by visit change in absolute neutrophil count (ANC) from baseline to post-treatment visits | Day 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85
Objective response rate (ORR) defined as the proportion of subjects with CR or PR as best overall response evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 on MRI or CT results | Day 1, 43, 85
Disease control rate (DCR) defined as the proportion of subjects with CR, PR, or SD as best overall response evaluated according to RECIST criteria version 1.1 on MRI or CT results | Day 1, 43, 85
Proportion of subjects with complete response (CR), partial response (PR), stable disease (SD), and progression disease (PD) as best overall response evaluated according to RECIST criteria version 1.1 on MRI or CT results | Day 1, 43, 85
Change in quality of life assessed by the Functional Assessment of Cancer Therapy Lung Cancer (FACT-L) total score from baseline to post-treatment visits | Day 1, 22, 43, 64, 85
  FACT-L total score ranges from 0 to 144. Higher values represent a worse outcome

IPD SHARING:
Plan to Share IPD: Undecided